CLINICAL TRIAL: NCT07343661
Title: Beyond Eosinophils: Proteomics to Identify Potential Biomarkers of Organ Damage and Response to MEPOLIZUMAB in EGPA
Brief Title: Beyond EOsinophils: proteoMICS to Identify Potential Biomarker of Organ Damage and Response to MEPOLIZUMAB in EGPA
Acronym: BEOMICS
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Azienda Ospedaliero Universitaria di Cagliari (Other)
Responsible Party: Principal Investigator, Giulia Costanzo, sub investigator, Azienda Ospedaliero Universitaria di Cagliari
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 14918-219771; GSK IIS Study 14918-219771 (Other Grant/Funding Number: GSK IIS)
Record Dates: First submitted 2025-09-25; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-11

CONDITIONS: EGPA - Eosinophilic Granulomatosis With Polyangiitis; Severe Asthma; Eosinophilic Asthma
Keywords: EGPA; severe asthma; eosinophilic asthma
MeSH Terms: conditions — Churg-Strauss Syndrome; Asthma; Pulmonary Eosinophilia | interventions — mepolizumab; Injections

STUDY DESIGN:
Intervention Model Description: According to the patients' groups evaluated in other publications with a robust statistical method and sample size calculation performed by the team, a sample of 90 patients can be considered sufficient to allow the realization of the study.
  The investigators plan to enroll 90 patients followed in Allergy and Clinical Immunology Centers divided into three groups:
  * 30 patients with EGPA with predominant ENT/asthmatic phenotype (longitudinal sampling before and after Mepolizumab treatment)
  * 30 patients with EGPA with vasculitic phenotype before and after immunosuppressive drugs (CYC, AZA, MTX) and/or Mepolizumab.
  * 30 patients with a diagnosis of severe eosinophilic asthma (longitudinal sampling before and after Mepolizumab treatment)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EGPA with predominant ENT/asthmatic phenotype (Experimental): Mepolizumab treatment
  Interventions: Drug: Mepolizumab 300 mg
- EGPA with vasculitic phenotype (Experimental): immunosuppressive drugs (CYC, AZA, MTX) and/or Mepolizumab
  Interventions: Drug: Mepolizumab 300 mg
- severe eosinophilic asthma (Active Comparator): before and after Mepolizumab treatment
  Interventions: Drug: Mepolizumab 100 MG Injection [Nucala]

INTERVENTIONS:
Drug: Mepolizumab 100 MG Injection [Nucala] — collect blood, salivary and sputum samples in both EGPA and severe asthmatic patients (as controls) at baseline and at different timepoints after starting treatment with mepolizumab, an anti-IL-5 drug, in order to cluster patients and to analyse the effect of the therapy during treatment and assess the disease progression on three key aspects of the disease: lung function and symptoms control, vasculitis and neuropathy.
  Arms: severe eosinophilic asthma
Drug: Mepolizumab 300 mg — collect blood, salivary and sputum samples in both EGPA and severe asthmatic patients (as controls) at baseline and at different timepoints after starting treatment with mepolizumab, an anti-IL-5 drug, in order to cluster patients and to analyse the effect of the therapy during treatment and assess the disease progression on three key aspects of the disease: lung function and symptoms control, vasculitis and neuropathy.
  Arms: EGPA with predominant ENT/asthmatic phenotype; EGPA with vasculitic phenotype

SUMMARY:
Aim of the study is to identify potential biomarkers, through a proteomic approach, which could be used to evaluate organ damage and predict the response to mepolizumab in a cohort of patients affected by EGPA. Proteomic analyses will be performed using a proteomic platform, based on a nano-HPLC- couplet to an high resolution ESI-MS device, on three types of biological matrices: blood, saliva and sputum samples in both EGPA and severe asthmatic patients (as controls) at baseline and at different time points after starting treatment with mepolizumab, an anti-IL-5 drug, in order to cluster patients and to analyze the effect of the therapy during treatment, assessing the disease progression on three key aspects: lung function and symptoms control, vasculitis and neuropathy. Plasma analysis will provide an overview of quantitative/qualitative proteomic variations at systemic level after drug administration; however, a less invasive procedure is often sufficient and would improve trial recruitment. On this regard, saliva is a biological fluid well suitable to be used in proteomic investigations for suggestion of potential disease biomarkers and includes various potential advantages compared with blood sample collection such as lower overall cost, lower infection risk, increased patient convenience, acceptability, compliance and uptake. Moreover, the protein composition of the human saliva includes both specific proteins of the oral cavity and proteins common to other tissues and bodily fluids, so saliva prognostic and diagnostic role is particularly interesting. Consequently, the plan is to compare the proteomic results of the non-invasive saliva testing to that of blood examination.

These data may be a further step to untangle the mechanisms of the disease and to characterize treatment's response, in the contest of a phenotype/endotype asthma management.

DETAILED DESCRIPTION:
The investigators plan to collect blood, salivary and sputum samples in both EGPA and severe asthmatic patients (as controls) at baseline and at different timepoints after starting treatment with mepolizumab, an anti-IL-5 drug, in order to cluster patients and to analyse the effect of the therapy during treatment and assess the disease progression on three key aspects of the disease: lung function and symptoms control, vasculitis and neuropathy.

untangle the mechanisms of the disease and to characterize response to treatment, in the context of a phenotype/endotype asthma and EGPA management.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent: Prior to start any study related activities, participants must be able and willing to provide written informed consent;
* Participants must have a current clinical diagnosis of asthma or EGPA;
* Physician decision to initiate treatment with mepolizumab.
* Patient has to be in treatment with medium-high dose ICS plus an additional controller in the least 6 months before screening and, if on OCS therapy, a stable dosage of prednisone (or equivalent dose of other steroids) in the 4 weeks before screening will be allowed. The above-indicated treatment has to be maintained by the patient all along the study.
* Adults aged 18 years or over.

Exclusion Criteria:

* Asthmatic patients receiving other biological treatment
* Participation in an interventional clinical trial in which the treatment regimen and/or monitoring is dictated by a protocol during the previous 12 months.
* Pregnant and breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-10-17 (Actual); Primary Completion 2026-10-17 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Saliva, sputum, and plasma proteomic profile of EGPA patients | From the data to the enrollment until the end of the study, up to 52 weeks.
  Obtain a proteomic profile of EGPA patients and severe asthmatic patients from blood, saliva and sputum.
  Analyse the samples after starting anti IL - 5 treatment ( mepolizumab ) and evaluate the possible disease modifying effect of the mepoliumab on vas

SECONDARY OUTCOMES:
If it is possible to predict the response to treatment by analyzing the proteomic profile of the patients. | From date of randomization until the date of first documented progression, assessed up to 24 months
  untangle the mechanisms of the disease and to characterize response to treatment, in the context of a phenotype/endotype asthma and EGPA management

CONTACTS AND LOCATIONS:
Overall Officials: STEFANO DEL GIACCO, MD, Principal Investigator — AZIENDA OSPEDALIERA UNIVERSITARIA CAGLIARI
Locations (1):
- Policlinico Duilio Casula AOU Cagliari, Cagliari, Cagliari, Italy

IPD SHARING:
Plan to Share IPD: No
PRIVACY

REFERENCES:
- [Background] Steinfeld J, Bradford ES, Brown J, Mallett S, Yancey SW, Akuthota P, Cid MC, Gleich GJ, Jayne D, Khoury P, Langford CA, Merkel PA, Moosig F, Specks U, Weller PF, Wechsler ME. Evaluation of clinical benefit from treatment with mepolizumab for patients with eosinophilic granulomatosis with polyangiitis. J Allergy Clin Immunol. 2019 Jun;143(6):2170-2177. doi: 10.1016/j.jaci.2018.11.041. Epub 2018 Dec 19. PMID 30578883
- [Background] Wechsler ME, Akuthota P, Jayne D, Khoury P, Klion A, Langford CA, Merkel PA, Moosig F, Specks U, Cid MC, Luqmani R, Brown J, Mallett S, Philipson R, Yancey SW, Steinfeld J, Weller PF, Gleich GJ; EGPA Mepolizumab Study Team. Mepolizumab or Placebo for Eosinophilic Granulomatosis with Polyangiitis. N Engl J Med. 2017 May 18;376(20):1921-1932. doi: 10.1056/NEJMoa1702079. PMID 28514601
- [Background] Kahn JE, Grandpeix-Guyodo C, Marroun I, Catherinot E, Mellot F, Roufosse F, Bletry O. Sustained response to mepolizumab in refractory Churg-Strauss syndrome. J Allergy Clin Immunol. 2010 Jan;125(1):267-70. doi: 10.1016/j.jaci.2009.10.014. No abstract available. PMID 20109753
- [Background] Puechal X, Pagnoux C, Baron G, Lifermann F, Geffray L, Quemeneur T, Saraux JL, Wislez M, Cottin V, Ruivard M, Limal N, Aouba A, Bonnotte B, Neel A, Agard C, Cohen P, Terrier B, Le Jeunne C, Mouthon L, Ravaud P, Guillevin L; French Vasculitis Study Group investigators. Non-severe eosinophilic granulomatosis with polyangiitis: long-term outcomes after remission-induction trial. Rheumatology (Oxford). 2019 Dec 1;58(12):2107-2116. doi: 10.1093/rheumatology/kez139. PMID 31056661
- [Background] Samson M, Puechal X, Devilliers H, Ribi C, Cohen P, Stern M, Pagnoux C, Mouthon L, Guillevin L; French Vasculitis Study Group. Long-term outcomes of 118 patients with eosinophilic granulomatosis with polyangiitis (Churg-Strauss syndrome) enrolled in two prospective trials. J Autoimmun. 2013 Jun;43:60-9. doi: 10.1016/j.jaut.2013.03.003. Epub 2013 Apr 13. PMID 23590801
- [Background] Jennette JC, Falk RJ, Bacon PA, Basu N, Cid MC, Ferrario F, Flores-Suarez LF, Gross WL, Guillevin L, Hagen EC, Hoffman GS, Jayne DR, Kallenberg CG, Lamprecht P, Langford CA, Luqmani RA, Mahr AD, Matteson EL, Merkel PA, Ozen S, Pusey CD, Rasmussen N, Rees AJ, Scott DG, Specks U, Stone JH, Takahashi K, Watts RA. 2012 revised International Chapel Hill Consensus Conference Nomenclature of Vasculitides. Arthritis Rheum. 2013 Jan;65(1):1-11. doi: 10.1002/art.37715. No abstract available. PMID 23045170

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan: revised protocol (2023-02-12): https://cdn.clinicaltrials.gov/large-docs/61/NCT07343661/Prot_SAP_000.pdf
  • Study Protocol: original (2023-02-12): https://cdn.clinicaltrials.gov/large-docs/61/NCT07343661/Prot_001.pdf
  • Study Protocol: COVER PAGE (2023-02-12): https://cdn.clinicaltrials.gov/large-docs/61/NCT07343661/Prot_002.pdf